CLINICAL TRIAL: NCT06608147
Title: Bone Marrow and Follicular Lymphoma
Brief Title: MOLyF : Bone Marrow and Follicular Lymphoma
Acronym: MOLyF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 35RC24_9716_MOLyF
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Lymphoma, Follicular
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Other: Sampling

INTERVENTIONS:
Other: Sampling — sternal bone marrow aspiration

SUMMARY:
This is a prospective single-center study designed to assess potential differences in cell composition between bone marrows of patients with follicular lymphoma and those from control subjects.

Follicular lymphoma is the most common indolent lymphoma. It is characterised by systematic relapses and bone marrow dissemination in 70% of patients at the time of diagnosis.

Although relapses are thought to be related to refractory tumour cells nested in a supportive microenvironment in the bone marrow, the mechanisms involved are poorly understood.

To study the specificities of the bone marrow of patients with follicular lymphoma, It is necessary to compare them with control samples.

This study takes advantage of surgeries involving sternotomies to recover lost bone marrow and establish a bone marrow bank of patients without hematological disease.

This bank will be used to set up control cohorts for other clinical trials involving patients with follicular lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient hospitalized in the thoracic, cardiac and vascular surgery department for surgery involving a sternotomy
* Patient with free, informed, written consent
* Patient covered by a health insurance scheme

Exclusion Criteria:

* History of haematological malignancy or haemogram disturbance
* Immunomodulating treatment: immunosuppressants, corticoids, antineoplastics
* Persons covered by articles L. 1121-5 to L. 1121-8 and L. 1122-1-2 of the French Public Health Code (e.g. minors, protected adults, etc.)].

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2034-10-01 (Estimated); Study Completion 2034-10-01 (Estimated)

PRIMARY OUTCOMES:
Flow cytometric quantification of cell populations | 1 day
  Bone marrow cell populations of lymphoma-free patients (lymphoid cells, myeloid cells, stromal cells and adventitial cells) will be quantified using a flow cytometry panel and compared with those of Follicular Lymphoma patients.

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Ferrant, MD, Study Chair — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided